CLINICAL TRIAL: NCT02713763
Title: Phase II Study to Evaluate Efficacy of Rechallenge With Sunitinib in Patients With Metastatic Pancreatic Neuroendocrine Tumor (pNETs) Well Differentiated G1/2 Advanced or Metastatic Who Previously Failed to Sunitinib.
Brief Title: Efficacy of Rechallenge With Sunitinib in Metastatic Pancreatic Neuroendocrine Tumor Previously Failed to Sunitinib
Acronym: RESUNET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Collaborators: Pfizer (Industry); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETNE-2016-01; 2015-005774-37 (EudraCT Number)
Record Dates: First submitted 2016-03-16; First posted 2016-03-21 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Pancreatic Neuroendocrine Tumour Metastatic
Keywords: Sunitinib
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sunitinib (Experimental): Sunitinib 37.5 mg/day
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib 37.5 mg/day
  Other Names: Sutent

SUMMARY:
The therapeutic goals in the management of pancreatic neuroendocrine tumors (pNET) are the control of symptoms and tumor growth control in order to improve patient survival.

In recent years, data from two phase III studies with targeted therapies, sunitinib and everolimus, have broadened the possibilities for treatment of patients with neuroendocrine tumors of the pancreas.

Unfortunately, patients progress and development of new active drugs and evaluating the best treatment approach is decisive.

Given the lack of data comparing the activity of different treatment strategies, final decisions are based on medical experience and consensus of experts. In this context, different questions are still unanswered, as which is the best sequence of treatment and if all patients can benefit from all available drugs.

Neuroendocrine pancreatic tumors are highly vascularized tumors in which cells may be dependent on this pathway for growth throughout the entire history of the tumor and in which inhibition of this pathway is crucial. On the other hand, this aspect has not been endorsed by the population of patients with pNET who have previously failed treatment with sunitinib.

In this scenario the investigators will assess retreatment with sunitinib to evaluate the activity of this drug in the context of therapeutic rescue in patients with metastatic pNET.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 18 years old and able to give their informed consent.
* Patients diagnosed with Neuroendocrine Tumor of pancreatic origin and histologically confirmed, G1/2 according to the World Health Organization (WHO) classification (Ki67 <20% and/or mitotic count >20 mitoses x 10 HPF).
* Metastatic disease progression in the 12 months prior to baseline visit documented by CT, MRI or Octreoscan.
* Progression to prior treatment with sunitinib administered for metastatic disease and have received at least 1 line and no more than 2 lines of subsequent systemic treatment.
* Measurable disease according to the following criteria RECIST version 1.1
* No disease that can be treated with surgery, radiotherapy or combined treatment with curative intent.
* Eastern Cooperative Oncology Group (ECOG) 0-2.
* Pretreatment with somatostatin analogues, chemotherapy, anti-VEGF (vascular endothelial growth factor) and mTOR (mammalian target of rapamycin) inhibitors prior to participation in the study is allowed.
* Adequately controlled blood pressure (BP) <150/90 mmHg.
* Hematologic Function: - Absolute neutrophil count >1500 / microliter (uL) - Platelets >100,000 / uL - Hemoglobin >5.6 mmol / L (9 g / dL)
* Liver function: total bilirubin < 1.5 x upper limit of normal (ULN), unless unconjugated hyperbilirubinemia or Gilbert syndrome. - Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5 x ULN (< 5 times in case of liver metastases).
* Renal function: calculated creatinine clearance according to Cockcroft-Gault > 30 ml / min.
* Blood coagulation: prothrombin time (PT) or International Normalized Ratio (INR) < 1.2 x ULN.
* Proteinuria <2+ urine dipstick. If > 2+ proteinuria, urinary protein <1 g / 24 h.
* Life expectancy> 3 months.
* Patient able to swallow the study drug and comply with the monitoring requirements of the study. - Women of childbearing potential must present a negative pregnancy test. Women of childbearing potential must agree to use contraception.
* Men whose partners are women of childbearing potential must use effective contraception.

Exclusion Criteria:

* Neuroendocrine tumors of pancreatic origin G3 according to WHO classification.
* Patients who received 3 or more lines of systemic treatment.
* Major surgery or trauma within 4 weeks prior to the first dose of sunitinib.
* Radiation therapy or tumor embolization within 2 weeks prior to the first dose of sunitinib.
* Chemotherapy, immunotherapy, biologic therapy or investigational therapy within the previous 2 weeks or 5 half-lives of the drug last received before the start of the first dose of sunitinib treatment.
* Prior treatment with high-dose chemotherapy that required hematopoietic rescue.
* Immunosuppressive therapy or prolonged treatment with corticosteroids concomitantly administered in the previous 3 months.
* Resolution to grade <2 (CTCAE according V4.03) of all previous related toxicities except alopecia treatments.
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 (according CTCAE V4.03) and/or that is progressing in severity, except alopecia.
* Treatment with potent inhibitors or inducers of CYP3A4 or known to prolong the QT interval in the previous 7 days.
* Prior radiotherapy to more than 25% of the bone marrow - Presence of uncontrolled metastatic brain disease, spinal cord compression, meningeal carcinomatosis or leptomeningeal disease.
* Any gastrointestinal malabsorption disorder or any other condition that, at investigator's criteria, may affect the absorption of sunitinib or increase the risk of bleeding or perforation.
* Presence of any non-healing wound or ulcer.
* Grade III/IV diarrhea in the screening period.
* Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri.
* Clinically significant cardio/cerebrovascular disease in the 6 months prior to treatment.
* Cardiac arrhythmias (NCI CTCAE version 4.0 grade >2), atrial fibrillation of any grade that requires medical treatment.
* Corrected QT interval (QTcF) > 180 msec.
* Active hemoptysis in the past 6 weeks.
* Evidence of active bleeding or bleeding diathesis.
* Presence of endobronchial lesions and/or lesions that infiltrate large vessels.
* Current treatment with acenocoumarol at therapeutic doses.
* Known HIV infection.
* Presence of uncontrolled active infection.
* Pregnant or breastfeeding women.
* Previous allergic reaction to components structurally similar to sunitinib or any of the excipients.
* Inability to discontinue any prohibited concomitant medication.
* Any illness (medical or psychiatric) or reason, in the investigator's opinion, that interferes with the patient's ability to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
6 months progression free survival | 6 months
  Time form start of treatment to progression disease

SECONDARY OUTCOMES:
Overall survival | 2 years
  Time form start of treatment to death
Progression free survival | 12 months
  Time form start of treatment to progression disease
Response duration | 12 months
  Time from first response to progression disease
Overall response rate | 12 months
  Complete response + partial response
Incidence of Adverse Events | 12 months
  Number of adverse events per patient

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Grande, Principal Investigator — MD Anderson Cancer Center MADRID
Locations (9):
- Spain (9):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Valle de Hebrón, Barcelona
  - Hospital Reina Sofía, Córdoba
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario J.M. Morales Meseguer, Murcia
  - Complejo Hospitalario Regional Virgen Del Rocío, Seville
  - Instituto Valenciano de Oncología, Valencia